CLINICAL TRIAL: NCT06662318
Title: Perioperative Analgesic Manipulations to Mitigate Pain After Elective Lumbar Spinal Surgeries: A Prospective Case-controlled Study
Brief Title: Perioperative Pain Management for Lumbar Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Azza Mahrous Shaffik, Clinical Lecturer of Anesthesia, Pain & ICU, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC 22/10/2024
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl; Dexmedetomidine; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group L (Active Comparator)
  Interventions: Drug: Lidocaine Hydrochloride
- Group D (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- Group F (Active Comparator)
  Interventions: Drug: Fentanyl Citrate

INTERVENTIONS:
Drug: Fentanyl Citrate — Fentanyl was given as a bolus of 1 µg/kg injected followed by a fentanyl infusion of 0.4 µg/kg/h. Fentanyl infusion was continued as Postoperative analgesia for 24 hours in a dose of 0.3 µg/kg/h.
  Arms: Group F
Drug: Dexmedetomidine — Dexmedetomidine was given as a loading dose of 0.6 µg/kg, which was diluted to a total volume of 10 cc of normal saline and injected before induction of anesthesia over 10 minutes. Then, a DXM infusion prepared to provide 0.2-0.7 µg/kg/h was started Intraoperative; Postoperative DXM infusion was provided in a dose of 0.15 µg/kg/h for 24-h.
  Arms: Group D
Drug: Lidocaine Hydrochloride — Lidocaine hydrochloride was provided as 2 mg/kg slowly IV before induction of anesthesia and as an IV infusion at a rate of 3 mg/kg/h. Postoprative lidocaine infusion at a dose of 1.5 mg/kg/h was administered for 24 Postoprative hours.
  Arms: Group L

SUMMARY:
Perioperative pain management is crucial for patients undergoing elective lumbar spine surgery. Moderate to severe postoperative pain can significantly impact recovery, worsen patient outcomes, and potentially lead to chronic pain.

Opioids have traditionally been the mainstay of postoperative pain management. However, their use is associated with several adverse effects, including nausea, vomiting, respiratory depression, and the risk of developing chronic pain. To mitigate these risks, there is a growing emphasis on multimodal analgesic approaches that combine various non-opioid medications to provide effective pain relief.

Non-opioid analgesics, such as nonsteroidal anti-inflammatory drugs (NSAIDs), regional anesthesia techniques, and adjuvant medications, can be used to reduce opioid requirements and improve patient outcomes. By carefully selecting and combining these modalities, clinicians can optimize pain management strategies for individual patients, minimizing the need for opioids and their associated side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had LDD and required lumbar discectomy,
* Patients are free of exclusion criteria and accepted to participate in the study.

Exclusion Criteria:

* The presence of other indications for spinal surgery;
* Obesity of grade ≥II;
* Patients of ASA grade >II;
* opioid dependence for preoperative pain;
* The presence of other causes of preoperative pain;
* The presence of preoperative psychiatric manifestations especially delirium and/or cognitive dysfunction;
* The presence of contraindications for the use of the study drugs;
* The presence of uncontrolled cardiac, renal, or hepatic disorders and essential hypertension.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reporting at least a 50% reduction in pain (measured by Numerical Rating Scale) in post-Operative Follow up for Lumbar Spine Surgery. | 2 months
  Value of non-opioid injection in Pain Reduction post operatively manifested by recurrence of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, El Qalyoubia, Egypt